CLINICAL TRIAL: NCT01453244
Title: Pharmacogenomic Research for Prediction of Drug Response in Korean Patients With Hepatitis C
Brief Title: Pharmacogenomic Research in Korean Patients With Hepatitis C
Status: Completed | Type: Observational
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Jae-Gook Shin, Jae-Gook Shin, Inje University
Other Study IDs: 11-037
Record Dates: First submitted 2011-10-13; First posted 2011-10-17 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; Pharmacogenomics; IL28B; ITPA
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — DNA extracted from blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SVR group: A patients who achieved SVR (sustained virologic response)
- non-SVR group: A patients who not achieved SVR (sustained virologic response)

SUMMARY:
The aim of this study is to investigate the relationships between drug response and the host genetic factors, viral factors and clinical factors in chronic hepatitis C patients (HCV). And thus, the investigators are trying to develop the pharmacogenomic guideline in the Korean patients with HCV.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C virus infected patients

Exclusion Criteria:

* Patients who infected Hepatitis B virus or Human immunodeficiency virus
* HCV infected patients previously treated with antiviral drugs
* Patients had a history of autoimmune hemolytic anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean patients with chronic hepatitis C
Sampling Method: Non-Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Sustained virological response (SVR) | 24 weeks after the end of treatment
  Undetectable HCV RNA in serum ( <15 IU/ml ) 24 weeks after the end of treatment

SECONDARY OUTCOMES:
Anemia | 4 weeks after start of treatment
  1. a reduction in Hemoglobin of >3.0 g/dL
  2. a reduction in Hemoglobin levels to 10.0g/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Gook Shin, M.D, phD, Principal Investigator — Inje University
Locations (1):
- Inje University, Busan, South Korea